CLINICAL TRIAL: NCT03512327
Title: Efficacy of the Autoimmune Protocol Diet for Inflammatory Bowel Disease
Brief Title: Autoimmune Protocol Diet and Inflammatory Bowel Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scripps Health (Other)
Responsible Party: Principal Investigator, Gauree G. Konijeti, Physician, Clinical Investigator, Scripps Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-6774
Record Dates: First submitted 2018-02-26; First posted 2018-04-30 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-12

CONDITIONS: Crohn Disease; Ulcerative Colitis; Inflammatory Bowel Diseases
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — aryl hydrocarbon receptor-interacting protein; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autoimmune protocol (AIP) diet (Experimental): Adult patients with active Crohn's disease or ulcerative colitis, undergoing 11 week autoimmune protocol diet, to examine therapeutic efficacy
  Interventions: Other: Autoimmune protocol (AIP) diet

INTERVENTIONS:
Other: Autoimmune protocol (AIP) diet — Autoimmune protocol diet, designed as a 6 week step wise elimination phase followed by 5 week maintenance phase.

SUMMARY:
There is limited data to guide the use of dietary change in the management of IBD, and it can prove challenging to implement in the setting of altered anatomy, comorbid conditions, and patient compliance. Therefore there is an important need to study diet as a therapy for IBD. Here, the investigators propose a novel study to evaluate the feasibility and efficacy of the autoimmune protocol (AIP) diet in patients with active Crohn's disease (CD) and ulcerative colitis (UC).

DETAILED DESCRIPTION:
The investigators propose a novel study to evaluate the feasibility and efficacy of the autoimmune paleo (AIP) diet in patients with Crohn's disease (CD) and ulcerative colitis (UC).

Specific aims:

1. To evaluate the effect of the AIP diet on clinical and endoscopic disease activity for CD and UC,
2. To examine changes in inflammatory biomarkers during AIP diet
3. To characterize changes in RNA expression from intestinal mucosal biopsy specimens from prior to diet initiation to end of the study.
4. To characterize changes in fecal microbiome during diet intervention

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. Able to provide written informed consent prior to screening and to comply with the requirements of the study protocol.
3. Established diagnosis of small bowel CD or colonic CD or ulcerative colitis
4. Confirmation of active CD or UC with recent (within 6 months of consent or prior to study start) objective evidence of endoscopically active disease on colonoscopy or computed tomography/magnetic resonance enterography or video capsule endoscopy
5. Any medications being currently used for IBD must remain stable during the study period with the exception of tapering of corticosteroids.
6. Current disease activity defined as a Harvey Bradshaw index ≥ 5 at baseline for CD or Partial Mayo Score ≥ 3 for UC
7. Established Facebook account
8. Comfortable with internet-based surveys and email

Exclusion Criteria:

1. If female, is pregnant or is breast feeding
2. Known celiac disease or subjects with a positive screen for celiac disease (elevated tissue transglutaminase antibodies)
3. Inability to provide informed consent or unwilling to participate
4. Evidence of untreated infection (e.g. Clostridium difficile)
5. Presence of stoma or J pouch
6. Bowel surgery within 12 weeks prior to enrollment and/or has surgery planned or deemed likely for inflammatory bowel disease during the study period
7. Use of tube or enteral feeding, elemental diet, or parenteral alimentation within 4 weeks prior to study initiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2016-12-10 (Actual); Study Completion 2016-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gauree G Konijeti, MD, MPH, Principal Investigator — Gastroenterologist, Clinical Investigator

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Autoimmune Protocol (AIP) Diet
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Autoimmune Protocol (AIP) Diet
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Remission for Crohn's Disease
Description: Clinical disease activity scores will be measured by Harvey Bradshaw Index for patients with Crohn's Disease (CD). The Harvey Bradshaw Index measures general well being, abdominal pain severity, number of stools daily, presence of abdominal mass, and complications. The Harvey Bradshaw Index ranges from 0-16, with lower values representing better outcome and higher values representing more disease activity. Clinical remission is defined as Harvey Bradshaw Index <5 for CD.
Time Frame: 11 weeks
Population: In this study, 9 out of the 15 participants had Crohn's disease. The other 6 participants had ulcerative colitis, so were not included in this subgroup analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Participants With Crohn's Disease: Adult patients with active Crohn's disease, undergoing 11 week autoimmune protocol diet, to examine therapeutic efficacy
Arm/Group | Participants With Crohn's Disease
Number analyzed (Participants) | 9
Participants | 6

2. Primary Outcome: Number of Participants With Clinical Remission for Ulcerative Colitis
Description: Clinical disease activity scores will be measured by Mayo score for patients with ulcerative colitis (UC). The Mayo score includes measures of stool frequency, rectal bleeding, physician global assessment, and endoscopic assessment. The Mayo score ranges from 0-12, with lower values representing better outcome and higher values representing more disease activity. Clinical remission is defined as Mayo score 2 or less for UC.
Time Frame: 11 weeks
Population: In this study, 6 out of the 15 participants had ulcerative colitis. The other 9 participants had Crohn's disease, so were not included in this subgroup analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Participants With Ulcerative Colitis: Adult patients with active ulcerative colitis, undergoing 11 week autoimmune protocol diet, to examine therapeutic efficacy
Arm/Group | Participants With Ulcerative Colitis
Number analyzed (Participants) | 6
Participants | 5

3. Secondary Outcome: Number of Participants With Mucosal Healing for Crohn's Disease or Ulcerative Colitis
Description: Number of participants with Crohn's disease or ulcerative colitis who have absence of erosions or ulcers on endoscopy or imaging
Time Frame: 11 weeks
Population: Of the 15 participants in this study, 7 had available followup endoscopic data available for assessment of mucosal healing.
Measure: Count of Participants; unit: Participants
Groups:
- Participants With Crohn's Disease or Ulcerative Colitis: Adult patients with active Crohn's disease or ulcerative colitis, undergoing 11 week autoimmune protocol diet, to examine therapeutic efficacy
  Autoimmune protocol (AIP) diet: Autoimmune protocol diet, designed as a 6 week step wise elimination phase followed by 5 week maintenance phase.
Arm/Group | Participants With Crohn's Disease or Ulcerative Colitis
Number analyzed (Participants) | 7
Participants | 7

4. Secondary Outcome: Changes in Inflammatory Biomarkers, Including C-reactive Protein (CRP), During Dietary Intervention
Description: Number of Participants with a change in C-reactive Protein Levels (inflammatory biomarker) from baseline to 11 weeks.
Time Frame: 11 weeks
Population: Of the 15 participants in this trial, 9 participants had available CRP data at the end of the study to evaluate changes in CRP.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Crohn's Disease or Ulcerative Colitis
Number analyzed (Participants) | 9
Participants | 9

5. Secondary Outcome: Changes in Inflammatory Biomarkers, Including Fecal Calprotectin (FC), During Dietary Intervention
Description: Number of Participants with a change in fecal calprotectin levels (inflammatory biomarker) from baseline to 11 weeks.
Time Frame: 11 weeks
Population: Of the 15 participants in the study, 6 patients had available fecal calprotectin data at 11 weeks for comparison
Measure: Count of Participants; unit: Participants
Groups:
- Patients With Crohn's Disease or Ulcerative Colitis: Adult patients with active Crohn's disease or ulcerative colitis, undergoing 11 week autoimmune protocol diet, to examine therapeutic efficacy
  Autoimmune protocol (AIP) diet: Autoimmune protocol diet, designed as a 6 week step wise elimination phase followed by 5 week maintenance phase.
Arm/Group | Patients With Crohn's Disease or Ulcerative Colitis
Number analyzed (Participants) | 6
Participants | 6

6. Secondary Outcome: Major Biological Processes Gene Ontology Terms Enriched in Downregulated and Upregulated Genes
Description: Description of changes in RNA expression from colonic biopsies from patients with ulcerative colitis from baseline to end of study (11 weeks). Specifically, examined top 10 major Biological Processes Gene Ontology Terms Enriched in Downregulated and Upregulated Genes
Time Frame: 11 weeks
Population: Outcome measure is descriptive. Of the 15 participants in this trial, 4 participants with ulcerative colitis had available colon biopsies at baseline and 11 weeks to examine changes in RNA expression in the colon. For all 4 participants, the 10 highest scoring Gene Ontology terms for biological processes associated with upregulated and downregulated genes were presented.
Measure: Number; unit: Enriched Gene Ontology Terms
Groups:
- Patients With Ulcerative Colitis: Adult patients with active ulcerative colitis, undergoing 11 week autoimmune protocol diet, to examine therapeutic efficacy
Arm/Group | Patients With Ulcerative Colitis
Number analyzed (Participants) | 4
Enriched Gene Ontology Terms | 10

7. Secondary Outcome: Changes in Fecal Microbiome Composition During Dietary Intervention
Description: Changes in fecal microbiome composition at baseline and at weeks 2, 4, 6, and 11 using 16S ribosomal RNA sequencing
Time Frame: 11 weeks
Population: Data was not collected. Fecal samples did not achieve quality control requirements in order to analyze data, so this substudy was terminated and analyses were not performed.
Arm/Group | Autoimmune Protocol (AIP) Diet
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Autoimmune Protocol (AIP) Diet
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 1/15
Other Adverse Events (participants affected / at risk) | 1/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Autoimmune Protocol (AIP) Diet (N=15)
Small bowel obstruction (Gastrointestinal disorders) | 1 (1) — Small bowel obstruction due to significant roughage intake
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Autoimmune Protocol (AIP) Diet (N=15)
Crohn's disease flare (Gastrointestinal disorders) | 1 (1) — Increase in gastrointestinal symptoms at week 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-01): https://cdn.clinicaltrials.gov/large-docs/27/NCT03512327/Prot_SAP_000.pdf